CLINICAL TRIAL: NCT03718208
Title: To Evaluate the Acceptability (Including Gastro Intestinal Tolerance and Compliance) of a Low Calorie Peptide Based Paediatric Tube-feed Formula; for Children Greater Than 1 Year of Age.
Brief Title: Acceptability and Tolerance Study of a Low Calorie Peptide Based Paediatric Tube Feed Formula.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Low calorie 001
Record Dates: First submitted 2018-08-22; First posted 2018-10-24 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2018-10

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paediatric formula (Experimental): Each child will receive for a period of seven days. The formula is a food for special medical purposes for use under medical supervision.
  The dietitian will determine the feeding regimen on an individual basis and the enteral formula will be provided via a feeding tube. One week intake diary, one week tolerance diary, product intake.
  Interventions: Dietary Supplement: Paediatric Formula

INTERVENTIONS:
Dietary Supplement: Paediatric Formula — Children will switch over to the low calorie paediatric feed. Intake diaries and tolerance diaries will be completed for one week.

SUMMARY:
This is an acceptability study to evaluate the gastrointestinal tolerance and compliance over a seven-day period, of a low calorie paediatric peptide based tube feed formula for the dietary management of participants with short bowel syndrome; intractable malabsorption; preoperative preparation of undernourished patients; inflammatory bowel disease; total gastrectomy; dysphagia; bowel fistulae;

The acceptability data from 15 participants will be collected in order to submit an application to the Advisory Committee on Borderline Substances (ACBS).

DETAILED DESCRIPTION:
Patients well established and stable on a standard or peptide enteral tube feed will be changed to a low calorie paediatric formula for a period of seven days. This group will act as their own controls. Each child will receive for a period of seven days the paediatric formula.

The dietitian will determine the feeding regimen on an individual basis and the enteral formula will be provided via a feeding tube. A baseline questionnaire will be completed by the dietitian to ensure eligibility of study, current stool patterns or symptoms and weight at the start of the study.

The parents will complete a week intake chart to monitor how much feed has been consumed each day and a tolerance diary to review gastrointestinal symptoms at the start and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Exclusively tube fed
* Paediatrics aged 1 year above who require a low calorie feed
* Children with Neurological impairment (NI) who require long term tube feeding
* Patients established on a standard or peptide Enteral formula (no gastrointestinal intolerances on a current formula)
* Willingly given, written, informed consent from patient or parent/guardian.
* Willingly given, written assent (if appropriate).

Exclusion Criteria:

* Inability to comply with the study protocol, in the opinion of the investigator
* Known food allergies to any ingredients (see ingredients list)
* Patients with significant renal or hepatic impairment
* Participation in another interventional study within 2 weeks of this study.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | Day 7 from baseline
  Incidence of gastrointestinal adverse effects [ Time Frame: day 7 from baseline ].
  Tolerance will be evaluated on the basis of the number of gastrointestinal events including diarrhea, constipation, bloating, distension, nausea, vomiting, burping, flatulence and regurgitation and abdominal discomfort or pain reported for subjects during their participation in the study.
  nausea, vomiting. burping, flatulence and regurgitation and abdominal discomfort or pain
Participant compliance | Day 7 from baseline
  Volume of test product prescribed versus actually taken

SECONDARY OUTCOMES:
Body weight | Day 7 from baseline
  Weight will be measured in Kg

CONTACTS AND LOCATIONS:
Overall Officials: Clare Thornton-Wood, BSc, Principal Investigator — Dietitian
Locations (3):
- United Kingdom (3):
  - Waldron Health Centre, Amersham
  - Alexandra Children's Hospital, Brighton
  - Gorton Clinic, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Yes see details below
Supporting Information: Study Protocol, CSR
Time Frame: The study has been published in a journal
Access Criteria: Avaliable on the internet
URL: https://www.heraldopenaccess.us/openaccess/tolerance-and-acceptability-of-a-low-calorie-paediatric-peptide-enteral-tube-formula-a-multicentre-trial-in-the-united-kingdom